CLINICAL TRIAL: NCT02436824
Title: A Phase II, Double-blind, Placebo-controlled, Randomized, Parallel-group Study to Determine the Safety and Efficacy of a Topical Patch (AB001) Following Daily Administration for 2 Weeks in Patients With Chronic Low Back Pain
Brief Title: A Study of a Topical Patch (AB001) in Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABS-201
Record Dates: First submitted 2015-04-30; First posted 2015-05-07 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Low Back Pain
Keywords: topical patch; chronic low back pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AB001 patch (Experimental): Two AB001 patches will be applied to the low back once daily for 14 days.
  Interventions: Drug: AB001 patch
- Placebo patch (Placebo Comparator): Identical in size and shape to the AB001 patch. Two placebo patches will be applied to the low back once daily for 14 days.
  Interventions: Other: Placebo patch

INTERVENTIONS:
Drug: AB001 patch — Two AB001 patches will be applied to the low back once daily for 14 days, the patches shall be removed after approximately 12 hours after daily application.
  Other Names: AB001
  Arms: AB001 patch
Other: Placebo patch — Two placebo patches will be applied to the low back once daily for 14 days, the patches shall be removed after approximately 12 hours after daily application.
  Arms: Placebo patch

SUMMARY:
The objectives of this study are to examine the safety, tolerability, and efficacy of repeated topical administration of AB001 topical patches for the treatment of chronic low back pain.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group study of the safety and efficacy of AB001 topical patches in patients with chronic low back pain. Subjects meeting inclusion criteria are randomized in a 1:1 ratio to receive AB001 patches or placebo patches. Two AB001 or placebo patches will be given topically once daily for 14 days. The primary end point is the change of low back pain intensity rated on a visual analog scale (VAS) scale on Day 15, the secondary end points include the subject global assessment (SGA) of low back pain, the subject global perceived effect (GPE) of study medication, the Roland-Morris Disability Questionnaire (RMDQ), and the pain assessment from subject diary (Days 1 - 3 only). Subjects' safety will be monitored throughout the study, including the adverse event (AE) incidence and severity, laboratory test results (hematology and clinical chemistry), vital signs, and physical examination.

ELIGIBILITY:
Inclusion Criteria:

1. Are generally healthy males or non-pregnant females, 18 to 75 years of age.
2. Have a body mass index (BMI) ≤35.
3. Have chronic low back pain for at least 3 months.
4. Have low back pain that is located inferior to the twelfth thoracic vertebra (T-12).
5. Back pain classified, using the Quebec Task Force system, as either Class 1 or Class 2.
6. Currently require use of analgesics for lower back pain (required at least 3 days per week for at least the last 4 weeks).
7. Have a score of 30 mm or greater on the visual analog scale (VAS) and a score of 2, 3, or 4 on the Subject Global Assessment (SGA) of Back Pain Scale at Screening.
8. Are willing to discontinue current analgesics for the 3 to 15 day washout period.
9. Have an increase of at least 10 mm or more from the score at Screening and an absolute score of 50 mm or more on the VAS (ie, VAS ≥ 50 mm) and a score of 3 or 4 on the SGA of Back Pain Scale at Baseline.
10. If female, are: 1).Of non-childbearing potential or have a confirmed clinical history of sterility or, 2).Of childbearing potential, must be willing to use effective contraception at trial entry and until completion.
11. Are willing to provide written informed consent.

Exclusion Criteria:

1. Have chronic lower back pain (CLBP) due to any of the following pathologies: infection, neoplasia, metabolic or structural disturbance of spine, lumbar radiculopathy, osteoporosis, hip dysplasia, inflammatory arthritis, ankylosing spondylitis, Paget's disease, cauda equine syndrome, gout, pseuodgout, fibromyalgia, post-surgical pain.
2. Have low back pain caused by major trauma.
3. Have excess hair, tattoo(s), or other dermatologic conditions in the patch application area that might interfere with efficacy evaluation.
4. Have had surgery for low back pain within the previous 6 months.
5. Have had clinical depression within 2 years or are currently undergoing treatment for depression;
6. Have a hypersensitivity to non-steroidal anti-inflammatory drugs (NSAIDs, including aspirin) or hypersensitivity to acetaminophen.
7. Have used opioids within 72 hours prior to the Baseline / Day 1 visit or during the course of the study.
8. Have used oral or injected corticosteroids chronically or intermittently within the past 60 days (oral), or 90 days (injected).
9. Are a current drug or alcohol abuser.
10. Are pregnant, plan to become pregnant during the study, or are breastfeeding.
11. Have a pending workman's compensation claim, litigation, or any other monetary settlement relating to the subject's lower back pain.
12. Have any chronic or acute medical condition that may pose a risk to the safety of the subject, or may interfere with the assessment of safety or efficacy in this trial.
13. Have a history of sensitivity to any component of the investigational product.
14. Have a known history of liver or kidney disorders (hepatic or renal insufficiency).
15. Have a known history of gastric ulcer, gastrointestinal bleeding, or significant cardiovascular events.
16. Have a history of cancer, other than treated basal cell carcinoma, within the past 5 years.
17. Use of any medication, including prescription, OTC, vitamins, herbal and/or mineral supplements, dietary supplements, enzyme altering agents within at least14 days prior to the first treatment or during the trial, which may influence the trial results.
18. Use of anti-coagulant medication within the past 30 days, including but not limited to heparins, warfarin/Coumadin, rivaroxaban/Xarelto, dabigatran/Pradaxa, apixaban/Eliquis, etc.
19. Participation in another clinical trial or received an investigational product within 30 days prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change of Pain intensity on VAS on Day 15 | From baseline to Day 15

SECONDARY OUTCOMES:
Change of Pain intensity on VAS on Day 8 | From baseline to Day 8
Change of Subject Global Assessment (SGA) of disease status/low back pain | From baseline to Day 8 and 15
Change of Roland-Morris Disability Questionnaire on low back pain | From baseline to Day 8 and 15
Subject Global Perceived Effect (GPE) of study medication | From baseline to Day 8 and 15
Pain Assessment from Subject Diaries | On Day 1 through Day 3
Safety Assessments on AEs | From baseline through Day 15
Safety Assessments on laboratory test | From baseline through Day 15
Safety Assessments on vital signs/physical examinations | From baseline through Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Changjin Wang, Study Director — Frontier Biotechnologies Inc.
Locations (9):
- United States (9):
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Pharma Research International, Inc., Naples, Florida
  - Georgia Institute for Clinical Research,LLC, Marietta, Georgia
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Atco Medical Associates, P.C., Atco, New Jersey
  - UniMed Center, East Brunswick, New Jersey
  - TKL Research, Inc., Fair Lawn, New Jersey
  - Upstate Clinical Trials, LLC, Spartanburg, South Carolina
  - Danville Orthopedic Clinic, Inc., Danville, Virginia